CLINICAL TRIAL: NCT01422291
Title: Pamukkale University Medical School,Dept. of Emergency Medicine
Brief Title: IV Paracetamol, Dexketoprofen or Morphine for the Treatment of Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Mustafa Serinken, Pamukkale University, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: serinken 002
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Low Back Pain
Keywords: Low back pain; paracetamol; dexketoprofen; morphine
MeSH Terms: conditions — Low Back Pain | interventions — Acetaminophen; Morphine; dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- morphine (Active Comparator)
  Interventions: Drug: Paracetamole
- Paracetamole, dexketoprofen (Experimental): Paracetamole, dexketoprofen
  Interventions: Drug: paracetamol; Drug: morphine; Drug: Dexketoprofen

INTERVENTIONS:
Drug: paracetamol — 1 gr
  Other Names: Perfalgan
  Arms: Paracetamole, dexketoprofen
Drug: morphine — 0.1mg/kg intravenous in 100 ml serum physiologic
  Other Names: Morphine CHL 0.01 gr
  Arms: Paracetamole, dexketoprofen
Drug: Dexketoprofen — 50 mg
  Other Names: Arveles
  Arms: Paracetamole, dexketoprofen
Drug: Paracetamole — 1 gr
  Other Names: Perfalgan
  Arms: morphine

SUMMARY:
This randomized, controlled trial evaluates the analgesic efficacy and safety of intravenous single-dose paracetamol, dexketoprofen and morphine for the treatment of low back pain.

DETAILED DESCRIPTION:
Study Design and Setting:

This is a single-center, prospective, randomized, double-blind, clinical trial performed in an ED of a tertiary care hospital with annual census of approximately 37.000 visits. The local ethics committee approved the study.

Interventions:

We conducted a randomized, controlled clinical trial comparing single intravenous doses of paracetamol (1 g), dexketoprofen (50 mg) and morphine (0.1 mg/kg) for patients presenting to the emergency department (ED) with suspected low back pain. Subjects with inadequate pain relief at 30 minutes received rescue fentanyl (0.75 microg/kg). We compared changes in pain intensity 30 minutes after treatment.

Methods of Measurements:

Subjects reported pain intensity on both a 100-mm visual analogue scale (limited by 'no pain' and 'the worst pain') and a 4-point verbal rating scale (no pain, mild, moderate, or severe pain) just before the drug administration, 15th minutes and 30th minutes after the study drug administration. The demographic features of study patients and adverse effects, nausea, vomiting, dizziness, vertigo, headache, hypotension, altered mental status, allergic reaction, itching, urinary retention, thoracic rigidity, respiratory depression and dry mouth, were recorded to the study form.

Outcome Measures The primary outcome measure was the pain reduction in VAS and VRS at 15th and 30th minutes. Secondary outcome measures were the need for rescue drug and the presence of any adverse event.

Primary Data Analysis:

The present study was planned as a superiority trial. When the 20 mm difference in VAS is accepted as clinically significant and the standard deviation is accepted as 25 mm, 35 patients are needed with each group with 95% power. All the analysis were implemented according to the intention to treat analysis. The precise of differences between time intervals within groups and between groups and statistical significance were expressed by 95% confidence intervals (95% CI).

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 16 to 55 years) with acute low back pain were eligible for inclusion in the study- -

Exclusion Criteria:

* Exclusion criteria included known allergy or contraindication to morphine, paracetamol,dexketoprofen or any opioid analgesic
* Hemodynamic instability
* Fever (temperature >38°C [100.4°F])
* Evidence of peritoneal inflammation
* Documented or suspected pregnancy
* Known or suspected aortic dissection or aneurysm, lombar disc hernia
* Use of any analgesic within 6 hours of ED presentation
* Previous study enrollment.
* Patients with known renal, pulmonary, cardiac, or hepatic failure, as well as those with renal transplantation, were also excluded.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Reduction in visual analogue scale | 15 minutes interval
  The pain of the study subjects was measured after 15th and 30th minutes later after the study drug administered

SECONDARY OUTCOMES:
Adverse events. | 30 minutes after
  30 minutes after the study drug administered